CLINICAL TRIAL: NCT06325306
Title: Physical Literacy-Based Intervention for Chronic Disease Management: A Quasi-Experimental Study Protocol
Brief Title: Physical Literacy-Based Intervention for Chronic Disease Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Alexandre MOUTON, Professor, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/392; B7072023000102 (Other: Comité d'Ethique Hospitalo-Facultaire Universitaire de Liège)
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Chronic Disease; Chronic Disease Management; Aging
Keywords: Physical literacy; Physical activity; Chronic Disease; quasi-experimental study; health promotion; group sessions
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants in this arm receive no specific intervention. They are on a waiting list for the 'Citoyen en mouvement pour ma santé' program, allowing for natural observation of their health progression without targeted physical literacy interventions. This group serves as a baseline to compare the effects of the adapted physical activity (APA) programs with and without physical literacy components.
- Traditional APA Group (Experimental): This group engages in a standard adapted physical activity program, focusing on improving physical fitness and mobility. The intervention is designed for chronic disease management, emphasizing regular physical exercises without an explicit incorporation of physical literacy principles. The same APA educator supervises all sessions to maintain consistency in the delivery of physical activity interventions.
  Interventions: Behavioral: Traditional APA
- APA+PL Group (Experimental): Participants in this arm participate in an adapted physical activity program enriched with physical literacy elements. The intervention aims to enhance physical activity engagement through increased motivation, confidence, knowledge, and understanding. This arm explores the added benefits of integrating physical literacy into traditional APA programs for chronic disease patients.
  Interventions: Behavioral: APA+PL

INTERVENTIONS:
Behavioral: Traditional APA — 12 sessions of 1,5 hour are organized (once per week). The first session is primarily focused on the PL assessment, followed by a comprehensive introduction to physical conditioning exercises. Each of the subsequent sessions (n=10), participants will receive an intervention focused on the development of their physical fitness (endurance, strength, flexibility, balance). Each session will commence with a 15 minute warm-up comprising of a blend of cardiovascular and joint mobilization exercises. The core part of each session will be dedicated to session-specific exercises targeting key physical competencies such as endurance, strength, flexibility, and balance, along with other motor skills. . The size of the group will never exceed a number of 15 participants. At the conclusion of each session, participants will be guided through a return-to-calm sequence that included stretching and relaxation exercises.
  Arms: Traditional APA Group
Behavioral: APA+PL — The general content and duration of this intervention is the same as in the traditional APA intervention, but with an extra particular and explicit emphasis on PL dimensions (6) during the sessions. While the dimension of physical competence is consistently incorporated into the sessions, the remaining 5 dimensions of PL are addressed twicely over the course of the semester with the setting of specific goals and intervention content. This could involve quizzes or games integrated into circuits or exercise workshops, role-play exercises simulating real-life situations, or social interactions between participants with a particular focus on PL-related topics. In addition to the sessions, a follow-up telephone call is scheduled between the educator and each participant during the 2 weeks following the initial PL assessment to share individual PL assessment results and assist participants in setting person-centered goals using a motivational interviewing technique.
  Arms: APA+PL Group

SUMMARY:
The goal of this quasi-experimental study is to evaluate the effectiveness of a physical literacy-based intervention for chronic disease management in adults with chronic diseases participating in adapted physical activity group sessions in Belgium. The main questions it aims to answer are:

* How does incorporating physical literacy elements in adapted physical activity sessions affect participants overall physical literacy levels?
* Can a physical literacy-oriented adapted physical activity program enhance long-term engagement in physical activities and improve health outcomes for chronic disease patients?

Participants will:

* Undergo assessments for physical literacy levels and health outcomes at the beginning, after three months, and at the end of the six-month period.
* Engage, in intervention groups, in adapted physical activity sessions, which may include physical fitness exercises and educational components on physical literacy.

Researchers will compare 3 groups: a control group, a traditional Adapted Physical Activity (APA) group, and a Physical Literacy Oriented APA (APA+PL) group to see if integrating physical literacy components results in improved physical literacy levels, better sustained engagement in physical activities, and enhanced health outcomes.

DETAILED DESCRIPTION:
The study employs a quasi-experimental design to investigate the impact of physical literacy-based interventions in chronic disease management. Participants are recruited from the Citoyen en mouvement pour ma santé program, designed for adults with chronic diseases in Belgium, facilitating their engagement in adapted physical activity (APA) group sessions. The study structure includes a control group (no intervention), a traditional APA group, and an APA with Physical Literacy (APA+PL) group, each consisting of approximately 65 participants to account for potential dropouts and ensure robust statistical analysis.

The intervention lasts six months, with initial and follow-up assessments at three and six months. These evaluations measure physical literacy dimensions-motivation, confidence, physical competence, knowledge, and engagement-using a combination of questionnaires and physical tests. The assessment tool, inspired by Whitehead's definitions and the IPLA framework, encompasses six core dimensions of physical literacy. It integrates closed-ended questions for quantitative analysis and open-ended questions for qualitative insights, offering a comprehensive view of participants physical literacy journey.

The APA+PL intervention is meticulously planned, following the Physical Literacy Interventions Reporting Template (PLIRT), focusing on enhancing physical literacy through tailored physical activity sessions. These sessions, led by qualified APA educators, are structured to integrate physical literacy elements seamlessly into the exercise routines. The program includes varied physical activities aiming to improve physical fitness (endurance, strength, flexibility, balance) and instill a deeper understanding and appreciation of physical literacy in participants.

The study data analysis plan involves a mixed-methods approach, capturing both the quantitative changes in physical literacy scores and the qualitative experiences of participants. Quantitative data will be analyzed using mixed ANOVA models to evaluate within-subject changes and between-group differences in physical literacy scores. Qualitative data, derived from open-ended questionnaire responses, will undergo thematic analysis to identify recurring themes and insights into the participants experiences and perceptions of the intervention.

Researchers will perform subgroup analyses based on age, gender, and chronic disease type, with adjusted analyses for potential confounders. The study seeks to understand the broader implications of physical literacy interventions in chronic disease management, aiming to inform future public health strategies and promote sustained engagement in physical activities among chronic disease patients.

This comprehensive approach to evaluating physical literacy interventions will contribute significantly to the understanding of how these interventions can be optimized to support chronic disease management in adult populations, potentially guiding future healthcare practices and policies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with one or more chronic diseases.
* Possessing a medical clearance to participate in physical activities.
* Enrolled in the Citoyen en mouvement pour ma santé program.
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Individuals younger than 18 years.
* Without a formal diagnosis of a chronic disease.
* Lacking medical clearance for engaging in physical activity.
* Not enrolled in the Citoyen en mouvement pour ma santé program.
* Unable to provide informed consent due to cognitive impairment or other reasons.
* Those who have severe mobility limitations or other health conditions that preclude safe participation in the physical activity sessions as determined by medical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Global Physical Literacy Score | Baseline, 3 months, and 6 months post-intervention
  The global physical literacy score is calculated based on the aggregated results from assessments covering six dimensions of physical literacy: motivation, confidence, physical competence, knowledge, engagement, and social interaction. Each dimension is scored out of a 8 points scale, and the total provides the global score (48 points), reflecting the comprehensive physical literacy level of participants: a higher score is associated with a higher physical literacy level.
Physical Activity Behavior and Engagement | Baseline, 3 months, and 6 months post-intervention
  This outcome measures the frequency, intensity, and regularity of physical activities performed by participants, assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-S). It quantifies physical activity in metabolic equivalent (MET) minutes per week, providing insight into the participants' engagement and adherence to physical activity routines. Score for PA behaviour/engagement relies on the IPAQ-S scoring protocol (low, moderate or high level of PA; /6 pts) and on the achievement of WHO recommendations for regular strength training activities (/2pts).
Motivation and Confidence in Physical Activity | Time Frame: Baseline, 3 months, and 6 months post-intervention
  Two closed-ended questions (Likert scale) related to motivation and confidence for the integration of regular physical activity in daily life are included, based on the preliminary tool assessment (Weerts & Mouton, 2023). Participants will also be asked to freely report (open-ended questions) their perceived facilitators and barriers to integrating physical activity into their daily lives. Scores for this dimension will be calculated according to level of answer given on the two closed-ended questions, on a 4-point likert scale (4pts per scale; a higher score is associated with a higher level).
Physical Competence | Baseline, 3 months, and 6 months post-intervention
  This outcome assesses the participants' abilities in physical tasks, including aerobic endurance, strength, flexibility, and balance. Tests like the 2-minute walk test, chair stand test, arm curl test, sit and reach test, and one-leg balance test are used to quantify physical competence, reflecting their functional fitness and physical literacy in this domain. The score for the physical competence will be based on the scoring scales used in our preliminary study (Mouton & Weerts, 2023), with 2pts attributed to each physical test (a higher score is associated with a higher level).
Knowledge and Understanding of Physical Activity | Baseline, 3 months, and 6 months post-intervention
  This outcome evaluates the participants awareness and comprehension of the principles and benefits of physical activity. Two closed-ended questions (likert-scale) ask the participant about their (1) perceived value of taking part in regular physical activity and (2) their perceived knowledge/understanding of main exercising guidelines (warm-up, progressiveness, and recovery) for health-related purposes. Finally, an open-ended question asked participants to write down what they know about WHO recommendations (2020) for aerobic PA. Scores for this dimension will be calculated according to level of answer given on the two closed-ended questions, on a 4-point likert scale (4pts per scale; a higher score is associated with a higher level).
Environment interactions | Baseline, 3 months, and 6 months post-intervention
  This outcome measures the extent of participants interaction and communication in physical activity contexts, assessing how social factors influence their engagement in physical activities. Two closed-ended questions (likert scale) are asked over the perceived support from peers (family, friends, etc.) for physical activity and over the perceived environmental (social and physical) opportunities for physical activity. Additionally, an open-ended question asks participants about the people and places that they would consider as helpful to help them to take part into a regular physical activity practice.. Scores for this dimension will be calculated according to level of answer given on the two closed-ended questions, on a 4-point likert scale (4pts per scale; a higher score is associated with a higher level).
Meaningful and Purposeful Activities | Baseline, 3 months, and 6 months post-intervention
  This dimension assesses how participants perceive the meaningfulness and purposefulness of physical activities in their lives. It examines the intrinsic value and emotional satisfaction derived from engaging in physical activities, highlighting the affective component of physical literacy. Two closed-ended questions (likert scale) ask participants about their perceived pleasure in taking part in physical activity, and about their perceptions of the meaningfulness/purposefulness of integrating physical activity in their daily life. Finally, participants are asked to describe in an open-ended question the characteristics of physical activities that they would personally consider as meaningful/purposeful. Scores for this dimension will be calculated according to level of answer given on the two closed ended-questions, on a 4-point likert scale (4pts per scale; a higher score is associated with a higher level).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Sportif du Sart-Tilman, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) that underlie the results reported in published articles, after deidentification, including text, tables, figures, and appendices. The shared data sets will encompass all collected IPD, such as demographic details, baseline characteristics, outcome measures, and intervention specifics. Access to these data will be provided upon request, following the publication of study results, to researchers who provide a methodologically sound proposal, with the aim of facilitating further research and understanding in the field of physical literacy and chronic disease management.
Supporting Information: Study Protocol, ICF
Time Frame: Time Frame: Beginning 3 months and ending 3 years after publication of results
  This time frame allows for the preparation of the dataset for sharing, ensuring data deidentification and compliance with privacy regulations, and gives a reasonable period for interested researchers to access and utilize the data for further research, while maintaining the relevance and timeliness of the data shared.
Access Criteria: Data sharing will be conditional upon the submission of a methodologically sound research proposal and a data sharing agreement to ensure the confidentiality and ethical use of the data. Proposals must detail the research questions, objectives, and statistical analysis plan. Requests will be reviewed by a committee comprising members of the original research team and external experts, ensuring that the proposed use of the data is scientifically valid and does not duplicate existing analyses. Approved researchers will be granted access to the data through a secure, online data-sharing platform. The data must be used solely for the approved research purposes and cannot be further shared without explicit permission.
URL: https://searchrxiv.org

REFERENCES:
- [Derived] Mouton A, Weerts JP, Carl J. Physical literacy-based intervention for chronic disease management: a quasi-experimental study protocol. BMC Sports Sci Med Rehabil. 2025 May 30;17(1):136. doi: 10.1186/s13102-025-01175-6. PMID 40448250
- See also: Website of the general project Citoyen en mouvement pour ma santé. — https://www.chuliege.be/jcms/c2_26224880/en-mouvement-pour-ma-sante/accueil

DOCUMENTS (1):
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT06325306/ICF_000.pdf